CLINICAL TRIAL: NCT01266200
Title: Identification of Cutaneous and Muscular Microcirculation and Inflammatory Response After Posterior Stabilization of the Spine
Brief Title: Identification of Microcirculation and Inflammation After Posterior Stabilization of the Spine
Acronym: MicroSpine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CTC-A10-027
Record Dates: First submitted 2010-12-17; First posted 2010-12-24 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Vertebral Fracture
Keywords: microcirculation; vertebral fracture; inflammation; minimal-invasive surgery
MeSH Terms: conditions — Spinal Fractures; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimal-invasive treatment (Mantis) (Active Comparator): Patients, who received a minimal-invasive surgery and the fracture was fixed by a system called Mantis
  Interventions: Procedure: Mantis; Procedure: XIA
- Conventional technique (XIA) (Active Comparator): Patients who received a surgical treatment including one long cut (conventional operation technique) and the fracture was fixed by a conventional system called XIA
  Interventions: Procedure: XIA

INTERVENTIONS:
Procedure: Mantis — percutaneous minimal-invasive technique at the thoracal-lumbal junction with for cuts of about 3 cms
  Other Names: minimalinvasive surgery of spine
  Arms: Minimal-invasive treatment (Mantis)
Procedure: XIA — Treatment of the fracture with Xia and conventional operation technique
  Other Names: open surgery of spine

SUMMARY:
In this project, with unstable vertebral fractures, the microcirculation of the skin and muscle (O2C,Laser-Doppler/White-light -Spectroscopy and contrast-enhanced sonography) will be evaluated in both conventional and in percutaneous minimally invasive technique (XIA versus Mantis) at the thoracolumbar junction.

DETAILED DESCRIPTION:
In this project, with unstable vertebral fractures, the microcirculation of the skin and muscle (O2C,Laser-Doppler/Whitelight-Spectroscopy and contrast-enhanced sonography) will be evaluated in both conventional and in percutaneous minimal-invasive technique (XIA versus Mantis) at the thoracolumbar junction. And after placing a fixator, the inflammatory potency (laboratory chemicals, cytokines, immune status) and the muscular injury (EMG) of acess are examined.

The study is planned as a randomized prospective study. In the study a total of at least 100 patients should be included, 50 with minimally invasive fixation-implantation and 50 patients with conventional procedure.

The radiological imaging (post-surgical control, possibly after mobilization, CT) ist routinely.

The patient outcome is determined using established scores (clinical score, visual analogue scale, SF-12).

The study also indicates by comparing the damage of the microcirculation of the two surgical techniques to make statements on wound healing and muscle blood flow heavily in order to filter out the less complications and tissue-method.

In this research project, the limits in the microcirculation measurement with the O2C and contrast enhanced sonography be established at an early stage to help in future wound healing disorders can be treated so well.

ELIGIBILITY:
Inclusion Criteria:

older than 18 years, fracture in thoracal-lumbal region, deceleration of agreement signed

Exclusion Criteria:

under age, pregnant, pathologic fractures, history of surgery in the examined area, history of metabolic bone disease, soft tissue damage, immunodeficient, polytrauma, history of significant heart or pulmonal diseases or diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Infection rate | 2 years
  Rate of postoperative wound edge necrosis and superficial or deep infection determined by wound redness, secretion of pus, detection of a microbial agens, CRP elevation and detection of fluid by sonography.

SECONDARY OUTCOMES:
Microcirculation, inflammation and functional clinical outcome | 2 years
  clinical (computer-assisted movement analysis, functional scores) and radiographic (Böhler angle, arthritis signs)control measure of cytokine level, microcirculatory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Knobe, MD, Principal Investigator — Dpt. of Orthopedic Trauma, RWTH Aachen University; Hans-Christoph Pape, MD, Study Chair — Dpt. of Orthopedic Trauma, RWTH Aachen University
Locations (1):
- RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany